CLINICAL TRIAL: NCT04456881
Title: Arthroscopic Clinical Study of Double Bundle Anatomical Reconstruction of Medial Patellofemoral Ligament
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014205
Record Dates: First submitted 2020-06-27; First posted 2020-07-07 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-01

CONDITIONS: Recurrent Patellar Dislocation
Keywords: arthroscopy; medial patellofemoral ligament
MeSH Terms: conditions — Patellar Dislocation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- anatomical reconstruction group of Patellofemoral ligament (Experimental)
  Interventions: Other: Patients with patellar dislocation undergo patellar femoral medial reconstruction

INTERVENTIONS:
Other: Patients with patellar dislocation undergo patellar femoral medial reconstruction — Arthroscopic double-beam anatomical reconstruction of medial patellofemoral ligament

SUMMARY:
Objective: To study the clinical effect of double-beam anatomical reconstruction of medial patellofemoral ligament under arthroscopy.

Methods: Double-beam anatomical reconstruction of medial patellofemoral ligament was performed under arthroscopy in patients admitted to our hospital for treatment of recurrent patellar dislocation. Carry out preoperative and postoperative evaluations, and conduct preoperative and postoperative comparative studies to clarify the clinical effect of the procedure.

Expected results: Arthroscopic double-beam anatomical reconstruction of the medial patellofemoral ligament can effectively restore the stability of the patella and the motor function of the knee joint.

Expected conclusion: Arthroscopic double-beam anatomical reconstruction of the medial patellofemoral ligament is an effective minimally invasive technique.

Keywords: knee joint; medial patellofemoral ligament; double-beam anatomical reconstruction; arthroscopy

ELIGIBILITY:
Inclusion Criteria:

* 17<age<60 years
* Recurrent patellar dislocation or instability

Exclusion Criteria:

- Bone spurs or bone protrusions on the D-type of the femoral pulley or proximal of the pulley.

Ages: 17 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2024-02-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
Lysholm score | 1 year after operation
  The Lysholm score consists of eight items including limping, locking, pain, stair climbing, use of supports, instability, swelling, and squatting. The higher values represent a better outcome.
International Knee Documentation Committee (IKDC) 2000 | 1 year after operation
  International Knee Documentation Committee (IKDC) 2000. The higher values represent a better outcome.
Tegner activity level score | 1 year after operation
  The highest level of activity that you participated in before your injury and the highest level you are able to participate in currently. The higher values represent a better outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Sports Medicine, Peking University Third Hospital, Beijing Key Laboratory of Sports Injuries， Beijing, China, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No